CLINICAL TRIAL: NCT01410669
Title: Is Motivational Interviewing an Effective Intervention for Women Coping With Intimate Partner Violence
Brief Title: Motivational Interviewing Intervention for Intimate Partner Violence
Acronym: ISIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Audrey F. Saftlas, MPH PhD, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 5R49CE000924-03 (NIH)
Record Dates: First submitted 2011-08-01; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Self-efficacy
Keywords: Self-efficacy; Intimate partner violence; Randomized clinical trial; Depression
MeSH Terms: conditions — Depression | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Motivational Interviewing (MI) (Experimental)
  Interventions: Behavioral: Motivational interviewing (MI)

INTERVENTIONS:
Behavioral: Motivational interviewing (MI) — MI is a "client-centered" counseling approach developed to deliver stage-tailored intervention messages using non-confrontational, supportive communication strategies. The client is encouraged to explore the barriers and facilitating factors associated with the behavior change. The interviewer's role is to guide the conversation and avoid use of conventional directive approaches (e.g., persuasion, providing information).
  In this trial, a trained motivational interviewer meets individually with patients randomized to the intervention for one-hour at baseline, followed by four MI telephone follow up contacts at 1-, 2-, and 4-months post baseline.

SUMMARY:
This project is a randomized trial to determine if motivational interviewing (MI) is an effective intervention to help women in abusive intimate relationships. The study objective is to motivate abused women to identify and achieve their own specific goals that can help them address the violence in their lives. This project will be integrated into the setting of a busy family planning clinic in the mid-western United States, which serves a largely rural population. Intimate partner violence (IPV) is screened using the Women's Experience with Battering Scale (WEB), a modified Abuse Assessment Screen (AAS), and the Danger Assessment Screen (DAS). An expected 250 women who screen positive for IPV will be enrolled, randomized to the intervention or to usual care group, and complete the 6-month study protocol. All subjects complete a self-administered computer-based questionnaire at the initial and 6-month follow up visits to measure self-efficacy (primary outcome), stage of readiness to change, selected IPV-related health correlates (e.g., depression), and steps taken and resources used. The MI intervention is an "active listening" counseling technique aimed at guiding the patient towards identifying feasible, personalized goals and steps she can take to increase her self-efficacy and control in the relationship. The trained study interviewer will work with participants to identify steps they can safely take and local resources to help them meet their goals. The MI protocol consists of a face-to-face counseling session at baseline with follow-up telephone interviews conducted at 1-, 2-, and 4-months post-intervention to reinforce the intervention and assess the participants' level safety. The control group will receive usual care, which includes talking with a Level 3 Domestic Violence Advocate and receiving a comprehensive list of domestic violence resources. Effectiveness of the MI intervention will be determined by increased self-efficacy, measured by the Domestic Violence Coping and Self-Efficacy Scale, a validated tool for use among women with a recent history of domestic abuse; and by a reduction in depressive symptoms (CESD-10). The impact of the intervention will be assessed by an increase in participants' readiness-to-change, and extent of their involvement in a wide variety of self-help and coping activities over the follow-up period. If successful, this screening and intervention program will be translated to other clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Screens positive for IPV
* Literate in either English or Spanish

Exclusion Criteria:

* Less than 18 years of age
* pregnant at time of screening and consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | Change from Baseline in Self efficacy at 6 months
  The Domestic Violence Coping Self-efficacy Measure by Benight et al (2004) was modified to measure self efficacy at baseline and 6-months post randomization

SECONDARY OUTCOMES:
Depression | Change from Baseline in depression at 6 months
  Depression at baseline and 6-month follow-up was measured using the 10 item Center for Epidemiologic Studies Depression Scale (CES-D )

CONTACTS AND LOCATIONS:
Overall Officials: Audrey F Saftlas, PhD, Principal Investigator — University of Iowa; Corinne Peek-Asa, PhD, Principal Investigator — University of Iowa
Locations (1):
- Iowa City, Iowa, United States

REFERENCES:
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505